CLINICAL TRIAL: NCT00140309
Title: TBTC Study 27: An Evaluation of the Activity and Tolerability of Moxifloxacin During the First Two Months of Treatment for Pulmonary Tuberculosis--A Double-Blind, Randomized, Multicenter Study by the Tuberculosis Trials Consortium
Brief Title: TBTC Study 27: Moxifloxacin vs Ethambutol for TB Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-3716
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Tuberculosis, Pulmonary
Keywords: TB; Pulmonary Tuberculosis; Tuberculosis; Pulmonary TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Moxifloxacin; Rifampin; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: moxifloxacin (with isoniazid, rifampin, pyrazinamide)

SUMMARY:
This study is a placebo-controlled factorial study, randomized to study drug (moxifloxacin vs. ethambutol) and treatment frequency (daily vs. thrice weekly after an initial two weeks of daily therapy) during the first two months of standard treatment (with isoniazid, rifampin, and pyrazinamide) for sputum smear-positive pulmonary tuberculosis.

DETAILED DESCRIPTION:
The primary objective of this Phase II clinical trial is to compare the safety and microbiological activity of a moxifloxacin-containing regimen (isoniazid, rifampin, pyrazinamide, moxifloxacin [HRZMoxi]) to a control regimen (isoniazid, rifampin, pyrazinamide, ethambutol [HRZE]) in the first two months of treatment of sputum smear-positive pulmonary tuberculosis. In addition, the study will evaluate whether intermittent administration (thrice-weekly after the first 2 weeks) of these regimens affects their tolerability and microbiological activity. The assessment of microbiological activity will be sputum culture-conversion. Improved sputum culture conversion after 2 months of treatment with a moxifloxacin-containing regimen would support phase 3 clinical trials of moxifloxacin in treatment regimens of less than the current 6 month standard regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected pulmonary tuberculosis with acid-fast bacilli in a stained sputum smear - patients whose sputum cultures do not grow M. tuberculosis and those having an M. tuberculosis isolate resistant to rifampin will be discontinued from the study, but followed for 14 days to detect late toxicities from study therapy. Patients having extra-pulmonary manifestations of tuberculosis, in addition to smear-positive pulmonary disease, are eligible for enrollment.
2. Willingness to have HIV testing performed, if HIV serostatus is not known or if the last documented negative HIV test was more than 6 months prior to enrollment
3. 7 or fewer days of tuberculosis therapy in the 6 months preceding enrollment
4. Age > 18 years
5. Karnofsky score of at least 60
6. Signed informed consent
7. Women with child-bearing potential must agree to practice an adequate (barrier) method of birth control or to abstain from heterosexual sex.
8. Laboratory parameters within 14 days of enrollment:

   * Serum amino aspartate transferase (AST) activity less than 3 times the upper limit of normal
   * Serum total bilirubin level less than 2.5 times upper limit of normal
   * Serum creatinine level less than 2 times upper limit of normal
   * Hemoglobin level of at least 7.0 g/dL
   * Platelet count of at least 50,000/mm3
   * Serum potassium > 3.0 meq/L
   * Negative pregnancy test (for women of childbearing potential)

Exclusion Criteria:

1. Breast-feeding
2. Known intolerance to any of the study drugs
3. Known allergy to any fluoroquinolone antibiotic
4. Current or planned therapy during the first 2 months of tuberculosis treatment using drugs having unacceptable interactions with rifampin (rifabutin can be substituted for rifampin during the continuation phase of therapy)
5. Current or planned antiretroviral therapy during the first 2 months of tuberculosis treatment
6. History of prolonged QT syndrome or current or planned therapy with quinidine, procainamide, amiodarone, sotalol, or ziprasidone during the first 2 months of tuberculosis treatment.
7. Pulmonary silicosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2003-07; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Two-month culture conversion
Serious Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: William Burman, MD, Principal Investigator — Denver Public Health Department; Richard E Chaisson, MD, Principal Investigator — Johns Hopkins University
Locations (23):
- United States (18):
  - University of Southern California Medical Center, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Denver Public Health Department, Denver, Colorado
  - Washington DC Veterans Administration Medical Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Hines Vetrans Administration Medical Center, Hines, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - New Jersey School of Medicine, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Harlem Hospital Center, New York, New York
  - Veterans Administration Tennessee Valley Health Care System, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston Veterans Administration Medical Center, Houston, Texas
  - Audie L Murphy Memorial Veterans Administration Medical Center, San Antonio, Texas
  - Seattle-King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute, Montreal, Quebec
- Nelson R Mandela School of Medicine, Durban, KwaZulu-Natal, South Africa
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- [Result] Burman WJ, Goldberg S, Johnson JL, Muzanye G, Engle M, Mosher AW, Choudhri S, Daley CL, Munsiff SS, Zhao Z, Vernon A, Chaisson RE. Moxifloxacin versus ethambutol in the first 2 months of treatment for pulmonary tuberculosis. Am J Respir Crit Care Med. 2006 Aug 1;174(3):331-8. doi: 10.1164/rccm.200603-360OC. Epub 2006 May 4. PMID 16675781
- [Derived] Zhang N, Savic RM, Boeree MJ, Peloquin CA, Weiner M, Heinrich N, Bliven-Sizemore E, Phillips PPJ, Hoelscher M, Whitworth W, Morlock G, Posey J, Stout JE, Mac Kenzie W, Aarnoutse R, Dooley KE; Tuberculosis Trials Consortium (TBTC) and Pan African Consortium for the Evaluation of Antituberculosis Antibiotics (PanACEA) Networks. Optimising pyrazinamide for the treatment of tuberculosis. Eur Respir J. 2021 Jul 20;58(1):2002013. doi: 10.1183/13993003.02013-2020. Print 2021 Jul. PMID 33542052
- See also: Tuberculosis Trials Consortium (TBTC) web page — http://www.cdc.gov/nchstp/tb/tbtc/default.htm